CLINICAL TRIAL: NCT00149669
Title: Employment-Based Addiction Pharmacotherapy
Brief Title: Employment-based Reinforcement of Naltrexone Ingestion and Abstinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00039284; R01DA019386 (NIH); NA_00039284 (Other: Johns Hopkins Medicine IRB)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2017-08-16 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-08

CONDITIONS: Cocaine-Related Disorders; Heroin Dependence; Opioid-Related Disorders; Substance Abuse, Intravenous
Keywords: Behavior Therapy; Cocaine; Cocaine (IV); Cocaine Abuse; Cocaine Dependence; Contingency management; HIV risk behaviors; Heroin; Naltrexone; Opioid Dependence; sexual risk behaviors
MeSH Terms: conditions — Cocaine-Related Disorders; Heroin Dependence; Opioid-Related Disorders; Substance Abuse, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Work Plus Naltrexone Prescription (No Intervention): Participants were prescribed naltrexone, but were not be required to ingest it to work. Participants could work and earn money, independent of whether or not they continued to take naltrexone.
- Work Plus Naltrexone Contingency (Experimental): Participants were required to ingest naltrexone to work, and received a brief pay decrease for missing a dose (employment-based reinforcement of naltrexone ingestion).
  Interventions: Behavioral: employment-based reinforcement

INTERVENTIONS:
Behavioral: employment-based reinforcement — Work Plus Naltrexone Contingency participants were required to ingest naltrexone to work, and received a brief pay decrease for missing a dose.
  Arms: Work Plus Naltrexone Contingency

SUMMARY:
A randomized study is planned over 5 years to evaluate the effectiveness of the Therapeutic Workplace in promoting naltrexone ingestion and abstinence in unemployed opiate-dependent injection drug users. Participants will be offered an opioid detoxification and naltrexone induction. Participants who complete the naltrexone induction will be randomly assigned to one of two groups. Both groups will be invited to work in the Therapeutic Workplace and prescribed naltrexone for 26 weeks. The groups will differ in the contingencies imposed to work and earn salary. Work Plus Naltrexone Contingency participants will be required to ingest naltrexone to work, and will receive a brief pay decrease for missing a dose. Work Plus Naltrexone Prescription participants will be prescribed naltrexone, but will not be required to ingest it to work. This study will provide a rigorous evaluation of a novel employment-based intervention, the Therapeutic Workplace, to promote naltrexone ingestion and drug abstinence in a population of injection drug users who are at considerable risk of spreading or contracting HIV infection. Hypotheses being tested in this study are: Naltrexone ingestion will be maintained in the group exposed to the employment-based naltrexone treatment significantly more than the group exposed to usual-care treatment package. Opiate abstinence will be maintained in the group exposed to the employment-based naltrexone treatment significantly more than the group exposed to usual-care treatment package.

DETAILED DESCRIPTION:
General Therapeutic Workplace Procedures The study was conducted in a model therapeutic workplace in which employment-based reinforcement contingencies are arranged to promote therapeutic behavior change. All participants were invited to attend the workplace for four hours every weekday to work on training programs that were almost fully automated. Participants earned vouchers that were exchangeable for goods and services in the community. Earnings were based on attendance in the workplace and performance in the training programs. Overall, voucher earnings were arranged such that participants could earn a base pay of $8.00/hour for the hours worked in the workplace plus approximately $2.00/hour for their performance on the training programs, for a total potential wage of $10/hour. Detailed descriptions of the therapeutic workplace, the web-based training programs, the staffing requirements, and the cost of the intervention can be found elsewhere. Participants in the Prescription group were eligible to work and earn vouchers independent of naltrexone consumption and/or drug use, however Contingency participants were only permitted to work when naltrexone consumption was objectively confirmed.

Assessment Procedures Assessments were conducted at study intake and every 30 days throughout the study. Primary assessment measures included the Addiction Severity Index-Lite to evaluate changes in medical, employment, alcohol, drug, social, legal and psychological functioning; the opiate, cocaine, alcohol and nicotine sections of the Composite International Diagnostic Interview to evaluate psychiatric disorders; the Risk Assessment of Behavior to evaluate HIV-risk behaviors; and the Beck Depression Inventory-II and Symptom Checklist-90 to evaluate psychosocial functioning. Additional measures were collected.

Naltrexone is contraindicated for patients with hepatic damage or reductions in liver functioning, and is rated in the FDA pregnancy category C. Therefore, blood samples were taken at intake, and months 1, 2, 3, and 5 for liver function (aminotransferase) levels, and pregnancy tests were conducted monthly. Naltrexone was discontinued permanently for one Contingency and one Prescription participant, and temporarily for one Contingency and one Prescription participant due to abnormal aminotransferase levels. Naltrexone was discontinued for one Contingency participant due to pregnancy.

Urine samples were collected under same-sex staff observation upon arrival to the workplace every Monday, Wednesday, and Friday and at each 30-day assessment. Urine samples were analyzed immediately onsite for evidence of opiates (morphine, >300ng/ml), and cocaine (benzoylecgonine, >300ng/ml) using an Abbott AxSYM® fluorescent polarization immunoassay system. Samples collected at 30-day assessments were also analyzed for evidence of buprenorphine, methadone, amphetamine, benzodiazepines, and naltrexone. Urine samples were analyzed for naltrexone using an Enzyme Linked Immunosorbent Assay (ELISA) procedure; values <5ng/ml were considered negative for naltrexone (Friends Laboratory, MD). Participants were informed of their urinalysis results but there were no consequences for positive test results.

Participants were instructed to notify study staff of any adverse events they experienced as soon as possible after the occurrence of the event. Any staff member who was notified by a participant of a potential adverse event filed a formal report into an automated system, which immediately distributed the reports to study investigators and key staff. Ongoing or unresolved adverse events were also included in a weekly adverse event report that was distributed to study investigators and key staff. At all 30-day assessments study staff assessed new adverse events and attempted to resolve any ongoing or unresolved adverse events. Participants were referred to medical staff to receive treatments and concomitant medications as needed, and reports were filed with the Institutional Review Board (IRB) and funding agency in accordance with the relevant institutional requirements and guidelines.

Oral Naltrexone Treatment Participants were required to complete opiate detoxification before being invited to attend the therapeutic workplace for induction onto oral naltrexone (Depade®; Mallinckrodt Inc.). All opiate detoxification and naltrexone inductions were overseen by a physician and were guided solely by clinical considerations. All participants were notified of the potential for heightened risk of overdose in relation to naltrexone treatment and after extended periods of opiate abstinence. These notifications were issued by study staff during the study consent process, and at monthly assessments, and were issued by medical staff prior to initiating naltrexone treatment, and whenever a blood draw was conducted. Overdose risk reminders were read aloud and signed by the study participants. Finally, monthly lunch-time overdose prevention seminars were provided and free pizza was provided to encourage seminar attendance.

During the 4-week induction period, participants were required to ingest scheduled doses of oral naltrexone to gain access to the therapeutic workplace. Induction onto oral naltrexone was determined by clinical judgment; participants were generally inducted using a 3-day dose run-up schedule (e.g., 12.5 mg, 25 mg, and 50 mg) in order to reach the full maintenance dose of 100 mg (Monday and Wednesday) and 150 mg (Friday) for the four-week period. Only participants who completed the induction period were considered eligible for randomization; these participants were invited to attend the therapeutic workplace for 26 weeks, and were offered oral naltrexone at no cost for the duration of the study. Participants were also offered access to outpatient drug abuse counseling that was provided independent of the workplace throughout their participation in the study.

Randomization Prior to group assignment, participants were stratified to an experimental group in a 1:1 ratio according to whether they attended the workplace on >85% of days during the 4-week induction period, provided >1 opiate positive urine sample during the final 2 weeks of the induction period, and provided >75% cocaine-positive urine samples during the 4-week induction period. Eligible participants were assigned to one of two experimental groups (i.e., Prescription or Contingency) using an urn randomization method that ensured all levels of each stratification variable were evenly distributed across the groups. This research design originally proposed three experimental groups; therefore, four participants were randomized into a third experimental group that required participants to ingest naltrexone under staff observation and provide an opiate and cocaine-negative urine sample to maintain maximum pay in the workplace. Due to logistical difficulties encountered early in the study, it became clear that it would not be possible to randomize a sample size large enough to support a 3-group comparison within the planned study duration. A second power analysis was completed to determine the appropriate sample size for a 2-group comparison (described below) and the third experimental group was eliminated. Data from participants randomized into the third group have not been included in these analyses.

Experimental Groups All participants were invited to attend the therapeutic workplace for 26 weeks. Prescription group participants were provided a take-home supply of oral naltrexone every 30 days and were allowed to access the workplace independent of naltrexone ingestion. Contingency participants were required to ingest oral naltrexone under staff observation every Monday, Wednesday, and Friday to gain access to the workplace. Contingency participants who missed a naltrexone dose were not permitted to access the workplace until they were able to resume naltrexone. Additionally, missing a scheduled dose resulted in a base pay reset from $8 per hour to $1 per hour. After a reset a participant's base pay increased by $1 per hour to a maximum of $8 per hour for every day that a participant attended the workplace for at least 5 minutes.

ELIGIBILITY:
Volunteers were eligible to participate if they

* were between the ages of 18 and 65 years,
* were unemployed (i.e., reporting no work in the past 30 days and earning $200 in taxable income per month),
* self-reported injection drug use and had visible track marks (assessed via visual inspection),
* provided a urine sample that tested positive for both opiates and cocaine upon entry into detoxification,
* met DSM-IV-TR criteria for opiate dependence,
* were medically approved to be maintained on naltrexone by the study physician,
* and lived within reasonable commuting distance to the research unit (i.e., in Baltimore City and the immediate surrounding area).

Volunteers were excluded if they

* had active hallucinations, delusions, or a thought disorder;
* were judged to be of imminent threat to harm self or others;
* were currently incarcerated, in a halfway house, or under constant monitoring;
* were pregnant or breastfeeding;
* had serum aminotransferase levels over 3 times normal;
* required opiates for other medical problems (and thus could not be maintained on naltrexone, which would block the effects on any opiate);
* reported an interest in methadone treatment;
* had active tuberculosis;
* or had physical limitations that would prevent typing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- The Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dunn KE, Defulio A, Everly JJ, Donlin WD, Aklin WM, Nuzzo PA, Leoutsakos JM, Umbricht A, Fingerhood M, Bigelow GE, Silverman K. Employment-based reinforcement of adherence to oral naltrexone treatment in unemployed injection drug users. Exp Clin Psychopharmacol. 2013 Feb;21(1):74-83. doi: 10.1037/a0030743. Epub 2012 Dec 3. PMID 23205722
- [Derived] Dunn K, DeFulio A, Everly JJ, Donlin WD, Aklin WM, Nuzzo PA, Leoutsakos JM, Umbricht A, Fingerhood M, Bigelow GE, Silverman K. Employment-based reinforcement of adherence to oral naltrexone in unemployed injection drug users: 12-month outcomes. Psychol Addict Behav. 2015 Jun;29(2):270-6. doi: 10.1037/adb0000010. Epub 2014 Aug 18. PMID 25134047

RESULTS

PARTICIPANT FLOW:
Groups:
- Work Plus Naltrexone Prescription; Work Plus Naltrexone Contingency: Participants who complete the naltrexone induction will be randomly assigned to one of two groups. Both groups will be invited to work in the Therapeutic Workplace and prescribed naltrexone for 26 weeks. The groups will differ in the contingencies imposed to work and earn salary. Work Plus Naltrexone Contingency participants will be required to ingest naltrexone to work, and will receive a brief pay decrease for missing a dose. Work Plus Naltrexone Prescription participants will be prescribed naltrexone, but will not be required to ingest it to work.
Period: Overall Study
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Started | 32 | 35
Completed | 29 | 30
Not Completed | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency | Total
Number analyzed (Participants) | 32 | 35 | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 35 | 67
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (7) | 43 (9) | 45 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 22 | 19 | 41
Region of Enrollment [Number; unit: participants]
  United States | 32 | 35 | 67

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Urine Samples Positive for Naltrexone
Description: The number of urine samples positive for naltrexone divided by the total number of urine samples times 100.
Time Frame: 6 months
Population: intent to treat
Measure: Mean (Full Range); unit: Percentage of Urine Samples
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 32 | 35
Percentage of Urine Samples | 21 [0 to 100] | 72 [0 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p < 0.01, General Estimating Equation (GEE); Odds Ratio (OR) = 8.67, 95% CI 2-sided [4.24 to 17.73]

2. Secondary Outcome: Percentage of Urine Samples Negative for Cocaine
Description: the number of urine samples that were negative for cocaine divided by the total number of urine samples) x 100
Time Frame: 6 months
Population: intent to treat
Measure: Mean (Full Range); unit: Percentage of Urine Samples
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 32 | 35
Percentage of Urine Samples | 53 [0 to 100] | 56 [0 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.82, General Estimating Equation (GEE); Odds Ratio (OR) = 0.91, 95% CI 2-sided [.43 to 1.95]

3. Secondary Outcome: Percentage of Urine Samples Negative for Opiates
Description: The number of urine samples negative for opiates divided by the total number of urine samples times 100.
Time Frame: 6 months
Population: intent to treat
Measure: Mean (Full Range); unit: Percentage of Urine Samples
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 32 | 35
Percentage of Urine Samples | 60 [0 to 100] | 71 [0 to 100]
Statistical Analysis 1: Comparison: Work Plus Naltrexone Prescription vs Work Plus Naltrexone Contingency; Test type: Superiority; p = 0.19, General Estimating Equation (GEE); Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.29 to 1.26]

4. Other Pre Specified Outcome: HIV Risk Behaviors
Description: Behaviors that place participants at risk for acquiring or transmitting HIV
Time Frame: 6 months
Population: These data were not analyzed due to limited funding. Funding this project has ended and we have no money to continue any summary or analyses.
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Cost Benefit Analysis
Description: The costs and economic benefits of the intervention
Time Frame: 6 months
Population: as for outcome 4
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Percentage of Urine/Breath Samples Negative for Other Drugs of Abuse
Description: The percentage of urine and breath samples that are negative for other drugs of abuse
Time Frame: 6 months
Population: as for outcome 4
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: Cocaine Positive Urine Samples
Description: The number of urine samples that were positive for cocaine
Time Frame: 6 months
Population: as for outcome 4
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Work Plus Naltrexone Prescription | Work Plus Naltrexone Contingency
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/35
Other Adverse Events (participants affected / at risk) | 4/32 | 7/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Work Plus Naltrexone Prescription (N=32) | Work Plus Naltrexone Contingency (N=35)
death by narcotic intoxication (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Work Plus Naltrexone Prescription (N=32) | Work Plus Naltrexone Contingency (N=35)
Ejaculation difficulty (Reproductive system and breast disorders) | 1 (1) | 2 (3)
General medical treatment, (General disorders) | 1 (1) | 0 (0)
Inpatient heroin detoxification (General disorders) | 1 (1) | 0 (0)
Jitters or shakes (General disorders) | 1 (1) | 0 (0)
Abnormal Liver Function Test (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting, diarrhea, chills (Gastrointestinal disorders) | 0 (0) | 1 (1)
E.R. for nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rapid heart rate (Cardiac disorders) | 0 (0) | 1 (1)
E.R. for adnominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
headache (General disorders) | 0 (0) | 1 (2)
Insomnia (General disorders) | 0 (0) | 1 (1)
Withdrawal (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No